CLINICAL TRIAL: NCT03031613
Title: Effects of Positive End Expiratory Pressure (PEEP) on Intracranial and Intraocular Pressure in Robot-assisted Laparoscopic Radical Prostatectomy
Brief Title: Effects of PEEP on Intracranial and Intraocular Pressure in Robot-assisted Laparoscopic Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3-2016-0263
Record Dates: First submitted 2017-01-05; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: intraocular pressure; intracerebral pressure
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEEP group (Experimental): Application of 5 cmH2O PEEP during mechanical ventilation
  Interventions: Procedure: PEEP group
- ZEEP group (Active Comparator): No application of PEEP during mechanical ventilation
  Interventions: Procedure: ZEEP group

INTERVENTIONS:
Procedure: PEEP group — Application of 5cmH20 positive end expiratory pressure
  Arms: PEEP group
Procedure: ZEEP group — No application of positive end expiratory pressure
  Arms: ZEEP group

SUMMARY:
To investigate the effects of positive end-expiratory pressure (PEEP) on the intracerebral pressure (ICP) and intraocular pressure (IOP) in patients undergoing robot assisted laparoscopic radical prostatectomy (RALRP)

DETAILED DESCRIPTION:
Application of PEEPmay reduce pulmonary complication following RALRP. Meanwhile, it may increase ICP and IOP, which has been debated for decades. Moreover, Trendelenburg position and pneumoperitoneum, which are mandatory for RALRP, may augment elevation of ICP and IOP. This study aims to investigate the effects of PEEP on the ICP and IOP in patients undergoing RALRP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotic-assisted laparoscopic radical prostatectomy

Exclusion Criteria:

* History of opthalmic disease or surgery
* History of brain disease or surgery
* Known ICP elevation
* Known IOP elevation
* Presence of lung bullae on chest x-ray
* History of pneumothorax

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
IOP | Changes from pre-induction (baseline) at Post-induction 5 min, Pneumoperitoneum insufflation and Trendelenburg position 5 min, Pneumoperitoneum insufflation and Trendelenburg position 30 min, Penumoperitoneum desufflation and supine position 5 min
  IOP is directly assessed by measurement of IOP with the Tono-Pen AVIA®
ICP | Changes from pre-induction (baseline) at Post-induction 5 min, Pneumoperitoneum insufflation and Trendelenburg position 5 min, Pneumoperitoneum insufflation and Trendelenburg position 30 min, Penumoperitoneum desufflation and supine position 5 min
  ICP is indirectly assessed by measurement of optic nerve sheath diameter(ONSD) with the ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Yonsei University Medical College Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No